CLINICAL TRIAL: NCT06002802
Title: Study on Biomarkers and Causative Factors of Complicated and/or Protracted Epstein-Barr Virus-associated Infectious Mononucleosis
Brief Title: Study on Infectious Mononucleosis in Munich
Acronym: IMMUC
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Collaborators: Helmholtz Zentrum München (Industry); German Cancer Research Center (Other); Ludwig-Maximilians - University of Munich (Other); Hannover Medical School (Other); University Hospital Freiburg (Other); German Center for Infection Research (Other)
Responsible Party: Sponsor
Other Study IDs: TTU 07.905/07.909
Record Dates: First submitted 2023-08-16; First posted 2023-08-21 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2023-08

CONDITIONS: Infectious Mononucleosis; Epstein-Barr Virus Infections
Keywords: EBV; Pfeiffer's glandular fever; Post-viral syndrome
MeSH Terms: conditions — Infectious Mononucleosis; Epstein-Barr Virus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, mouthwashes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational clinical study aims at the identification of novel biomarkers and causative factors of complicated and/or protracted Epstein-Barr virus-associated infectious mononucleosis (IM).

Clinical, biochemical, and routine virological data were collected from 200 patients with IM, novel analytical tools were implemented, and immunological and virological experimental data were generated using blood samples and mouthwashes. Patients have been investigated within four weeks after the onset of symptoms as well as one month and six months thereafter.

DETAILED DESCRIPTION:
EBV-associated diseases are a severe and global health problem, and novel tools and targets for a better pathogenetic understanding, diagnosis, treatment, and prevention are clearly needed. Here we propose to use several novel experimental approaches to investigate immunological, virological, biochemical, and clinical features in an observational study on Munich IM patients.

This study aims at identifying biomarkers and causative factors of protracted and/or complicated IM to facilitate the development of novel approaches to early diagnosis, therapy, and prevention of severe, life-threatening, and chronic EBV-associated diseases, including post-viral syndromes.

Two hundred patients with IM onset within the last four weeks were recruited from Munich health care institutions and were re-investigated at one and six months after the onset of symptoms. A novel diagnostic scoring system was developed to indicate the severity, complexity, and protraction of symptoms.

Investigated clinical parameters, including reported symptoms and physical signs of IM, as well as candidate risk factors in the medical history of patients and family members. Peripheral blood was analysed by established and novel analytical assays to determine the immunological and virological phenotypes of IM, and viral load was determined in mouthwashes.

ELIGIBILITY:
Inclusion Criteria:

* IM onset within the last four weeks
* with at least one of four typical clinical findings (tonsillopharyngitis, fever, lymphadenopathy, fatigue) - virological findings indicating primary EBV infection (EBV-specific antibodies, EBV DNA).

Exclusion Criteria:

* Pregnancy
* transfusion
* and/or transplantation during the last year
* and/or no informed consent.

Ages: 0 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 200 patients with infectious mononucleosis.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Severity | Six months
  Maximal severity of symptoms during the course of IM according the the IMMUC-Score.
Complexity | Six months
  Maximal complexity of symptoms during the course of IM according the the IMMUC-Score
Protraction | Six months
  Maximal protraction of symptoms during the course of IM according the the IMMUC-Score.

SECONDARY OUTCOMES:
Immune status | Within four weeks post symptom onset and at one and six months thereafter.
  Cellular and humoral immune status, EBV viral load, antibodies against EBV proteome.

CONTACTS AND LOCATIONS:
Locations (1):
- MRI Chonic Fatigue Center for Young People (MCFC), Children's Hospital, Technical University of Munich & Munich Municipal Hospital, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Federal Ministry of Education and Research — https://www.gesundheitsforschung-bmbf.de/de/epstein-barr-virus-von-harmlos-bis-folgenschwer-7238.php
- See also: German Center for Infection Research — https://www.dzif.de/en/epstein-barr-virus-harmless-severe-consequences